CLINICAL TRIAL: NCT02508545
Title: Influence of Gravity on the Perception of Egocentric Distance (Blindpulling)
Acronym: Blindpulling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-002
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- perceived egocentric distance measurements - parabolic flight (Other): perceived egocentric distance (PED) measurements during parabolic flight
  Interventions: Other: perceived egocentric distance (PED) measurements; Other: Parabolic flight

INTERVENTIONS:
Other: perceived egocentric distance (PED) measurements
Other: Parabolic flight

SUMMARY:
Parabolic flight is the only ground-based condition in which weightlessness (0G) can be created long enough for safely testing changes in human perception and behavior. In addition to the 0G period, parabolic flight generates equal duration periods of 1.8G, which present another unique opportunity to test the same responses to hypergravity and back to 1G.

Cognitive function, together with good oculomotor control, eye-hand coordination, and spatial orientation perception, is a critical subsystem that is used by the CNS in the control of vehicles and other complex systems in a high-level integrative function. Evidence from space flight research demonstrates that the function of each of these subsystems is altered by the transitions in gravito-inertial force levels. These neuro-vestibular alterations, unfortunately, correspond to mission phases where physical and cognitive performance are particularly critical for crew safety and mission success. To date, there is only limited operational evidence that these alterations cause functional impacts on mission-critical vehicle (or complex system) control capabilities. However, the true operational risks will be estimable only after the investigators have filled the knowledge gaps and when the investigators can accurately assess integrated performance in off-nominal operational settings.

Accurate perception of self-in-space motion and self-motion relative to other objects are critical to piloting, driving, and remote manipulator operations. Immediately after space flight, most crewmembers have reported some degree of disorientation/perceptual illusion, often accompanied by nausea (or other symptoms of motion sickness), and frequently manifested by lack of coordination, particularly during locomotion. Despite recent, intensive training, some Shuttle landings were outside of the desired performance boundaries. Scores indicating neurovestibular dysfunction in returning astronauts generally correlated with poorer flying performances, including a lower approach and landing shorter, faster, and harder. An underestimation of distance, coupled to an overestimation of tilt magnitude or misperception of the type of motion, could be at the origin of these poorer performances.

This study should confirm that the unloading of the otoliths in weightlessness induces an alteration in the egocentric reference during space flight. Errors in egocentric localization might contribute at a higher level to the computation of misleading world-centered representations, and therefore be partly responsible for illusory sensations and motion sickness symptoms during space flight, and postural instability and oscillopsia after returning in a reduced or terrestrial gravitational force level.

Beside their fundamental implications, the results of this study have also practical implications in the design of man-machine interfaces. Changes in judgment of distance in microgravity or in reduced gravity affect crew posture and reach, display orientation, and other visual cues, which should be considered in hardware and operations design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 21 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with medical history of oculomotor disorders
* Person with medical history of vestibular disorders
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Blind pulling error, i.e. difference between the actual position of the visual target and the final position of the subject between 1G, 1.8G, and 0G during parabolic flight and with blind pulling evaluation method | baseline
Blind pulling error, i.e. difference between the actual position of the visual target and the final position of the subject between 1G, 1.8G, and 0G during parabolic flight and with verbal report evaluation method | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France